CLINICAL TRIAL: NCT00138346
Title: Epidemiology of Human Cystic Hydatid Disease
Brief Title: Epi Cystic Hydatid Disease Peru
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 04-045
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2006-12

CONDITIONS: E. Granulosus Cystic Hydatid d
Keywords: hydatid disease, Echinococcus granulosus, tapeworm
MeSH Terms: conditions — Echinococcosis; Cestode Infections

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This is a study developed by researchers from the Universidad Peruana Cayetano Heredia, the Universidad Mayor de San Marcos and other local and foreign institutions. Researchers are performing this research in human beings and animals, in order to determine the best way to understand and eliminate a parasite called Echinococcus granulosus (tapeworm). The parasite grows and develops in the dogs´ bowel. The tapeworm produces eggs which are eliminated among the feces and remain in the environment. Individuals may accidentally ingest the eggs through contaminated food or drinks and develop a disease called cystic hydatid disease. This disease mainly affects the human lungs and liver. The parasite grows in the shape of a water bag and it can jeopardize human life. It also affects sheep, goats, llamas and alpacas. The study will enroll almost 840 volunteers who are older than 5 years of age. It will last about 3 years.

DETAILED DESCRIPTION:
This is a 3 year study of approximately 840 male and female subjects aged 5 years old and above to be conducted in a Peruvian Highland community in Lima, Peru in order to described the dynamic and associated risk factors to both human infection and Cystic Hydatid Disease (CHD). The purpose is to determine the prevalence and incidence of both infection and disease in human population, to assess the proportion of seroconversion (positive to negative) through follow-up of the same indiviuals every year and to identify risk factors related to human infection and disease by using baseline questionnaire (e.g. husbandry practices and education level). Echinococcal infection is prevalent in regions of the world where dogs are used to care for large herds (Lima, Peru). This study involves collection of 5 ml of blood every year for 3 years. In addition, CXR and abdominal US will also be performed. Signs and symptoms of hydatid disease depend on the organ involved (lungs and liver) and the size of the cyst. At this time, the best therapeutic approach is surgical intervention preceded by careful radiological evaluation plus adjuvant chemotherapy. The mortality rate post surgery is 1-4% and for those patients who refuse to have surgery, 60%. Despite the presence of current methods of control, the parasite prevalence appears to be increasing worldwide therefore this study will obtain data to implement a control program to eradicate this zoonosis.

ELIGIBILITY:
Inclusion Criteria:

1. Living in study area (Cooperative Tupac Amaru).
2. Older than five-years old

Exclusion Criteria:

1. Pregnant woman (only for chest X-ray procedure).

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 840
Dates: Start 2004-08; Study Completion 2007-04

CONTACTS AND LOCATIONS:
Locations (2):
- Peru (2):
  - Universidad Nacional Mayor de San Marcos, Lima
  - Universidad Peruana Cayetano Heredia, Lima